CLINICAL TRIAL: NCT05447624
Title: The Effect of Radiofrequency Ablation on the Results of the Genicular Nerve Number in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 092021654
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Knee; Radiofrequency Ablation; Genicular Nerve
Keywords: Osteoarthritis Knee; Genicular Nerve; Radiofrequency Ablation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing ablation of two of the genicular nerve branches (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation of genicular nerves
- Patients undergoing ablation of three of the genicular nerve branches (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation of genicular nerves

INTERVENTIONS:
Procedure: Radiofrequency ablation of genicular nerves — The RF cannula will be placed near the nerve with an in-plane technique from proximal to distal. Sensory stimulation will be performed at 50 Hz to ensure localization. The sensory threshold should be less than 0.6 V. To prevent ablation of the motor nerves, when the nerve is stimulated with 2.0 V at 2 Hz, it will be seen that there is no fasciculation in the relevant region of the lower extremity. Before starting the ablation procedure, 2 mL of 1% lidocaine solution will be injected around the nerve, after vascularity control, in order to reduce the pain and the risk of neuritis during the procedure. Then the temperature will be adjusted to 80° degrees and applied for 90 seconds and the process will be terminated.

SUMMARY:
Knee osteoarthritis is a disease that increases in frequency with age and decreases the quality of life and physical activity by leading to a decrease in pain and joint range of motion. Basically, the articular cartilage is affected and clinically pain, joint stiffness, crepitation and effusion are seen. In imaging techniques applied with weight-bearing, varying degrees of joint narrowing are observed, although it is more common in the medial. Treatment options include conservative approaches such as weight loss, physical therapy, analgesics, or invasive approaches such as intra-articular injections, peripheral nerve blocks, joint-sparing surgery or total knee replacement. Surgical operation should be considered in the treatment when conservative treatments are insufficient. However, the advanced age of this patient group and the large number of comorbidities reduce the possibility of surgical operation. Although treatment cannot be cured in knee osteoarthritis, the aim of the treatment is to decrease the pain, increase the patient's quality of life and physical capacity, and slow down the progression of the disease.

Although the radiofrequency ablation (RFA) technique has been used since the 1970s, the first application area was trigeminal neuralgia. Later, its use in neck and back pain became widespread, but the first randomized controlled study on its use in knee osteoarthritis was Choi et al. Made by in 2011. The purpose of radiofrequency ablation applied to the genicular nerves that receive the sensation of the knee joint capsule is to prevent sensory transmission and reduce the sensation of pain by creating axonal damage to these nerves. Since the use of RFA in knee osteoarthritis is relatively new, studies on the development of the technique continue. Fluoroscopy device or ultrasonography can be used as imaging method to show target nerves or to place the RFA electrode in the correct localization.

The investigators hypothesis; based on the more prominent medial involvement in knee osteoarthritis, the conventional RFA procedure applied to the 3 genicular nerves (SMGN, IMGN, SLGN) is not superior to the RFA procedure applied to the medial SMGN and IMGN branches.

ELIGIBILITY:
Inclusion Criteria:

* Be over 50 years old and under 80 years old
* Symptom duration is at least 3 months
* Pre-procedure NRS score of more than 6
* Kellgren-Lawrence stage 3-4
* Failure to respond to conservative treatments
* Having given consent to participate in the study
* The patient's ability to speak and read and write Turkish

Exclusion Criteria:

* Body mass index of 41 kg/m2 or more
* Acute knee injury
* Chronic pain syndrome (fibromyalgia syndrome, chronic fatigue syndrome, etc.)
* Lumbar radicular pain
* Uncontrolled diabetes mellitus
* Presence of bleeding diathesis
* Hemodynamic instability
* Pacemaker presence
* History of septic arthritis or active local or systemic infection
* Having a history of surgery on the knee to be treated
* Intra-articular injection of the knee within 3 months
* Cognitive impairment
* Presence of genu valgus deformity
* Presence of secondary knee osteoarthritis (due to trauma, rheumatoid arthritis, systemic inflammatory diseases such as gout, kinetic chain disorder due to congenital hip dislocation)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 3 months
  It is a scale on which patients score their pain between 0 and 10, with 0 = "no pain" and 10 = "worst pain imaginable"

SECONDARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | 3 months
  WOMAC is a 24-item scale under the headings of pain, stiffness and functional activity. Patients rate the amount of strain, pain felt, and joint stiffness during daily activities between 0 and 4 (0 is the best, 4 is the worst), and the total score is between 0 and 96.
SF-36 (Short Form-36) | 3 months
  SF-36 is a scale in which 8 sub-parameters such as physical function, body pain, and emotional well-being are evaluated with 36 questions.
TUG (Timed Up and Go Test) | 3 months
  In the TUG test, the patient gets up from the chair with the command of the person performing the test, and after pressing the line drawn 3 meters on the floor with both feet before, he returns and sits on the chair. The tester measures the time elapsed between the stand up command and the patient's back contacting the chair. The patient can get support from the chair while getting up and sitting, and can rest whenever he wants, provided that he does not sit. During the test, the patient walks in the shoes he always uses and at his daily walking speed.
use of analgesic drugs | 3 months
  During the follow-up period, the analgesic drugs used by the patients, if any, and the information about the use of these drugs during the follow-up period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No